CLINICAL TRIAL: NCT00839774
Title: Effect of Pulse Fractions on Indices of Lipid, Carbohydrate and Energy Metabolism as Well as Oxidative Status in Overweight, Hyperlipidemic Individuals
Brief Title: Effect of Pulse Fractions on Indices on Cardiovascular Disease and Diabetes Risk Factors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Pulse Canada (Other)
Responsible Party: Dr. Peter J.H. Jones/ Director of the Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: B2006:129
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2008-08

CONDITIONS: Cardiovascular Disease
Keywords: Peas; Cardiovascular; Diabetes; Insulin; Insulin resistance; Abdominal fat
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Whole yellow pea flour
  Interventions: Other: Whole yellow pea flour
- 2 (Experimental): Fractionated yellow pea flour
  Interventions: Other: Fractionated pea flour
- 3 (Experimental): White wheat flour
  Interventions: Other: White wheat flour

INTERVENTIONS:
Other: Whole yellow pea flour — Whole pea flour was administered at 50 g/day.
  Arms: 1
Other: Fractionated pea flour — Fractionated pea flour was administered according to the level of fiber in whole pea flour treatment. 12 g/day
  Arms: 2
Other: White wheat flour — White wheat flour will be administered at 50 g/day
  Arms: 3

SUMMARY:
The purpose of this study is to determine if whole and fractionated yellow pea flour, administered at USDA recommended dosages (50 g/day), improve risk factors associated with cardiovascular disease and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 40 kg/m2
* Hypercholesterolemic

Exclusion Criteria:

* Smoking
* Use of prescription and natural lipid lowering therapies
* Myocardial infarction
* Coronary artery bypass
* Angina
* Congestive heart failure,
* Inflammatory bowel disease
* Pancreatitis
* Renal disease
* Diabetes
* Chronic alcohol usage (> 2 drinks/day).
* Cancer
* Eating disorders
* Expending > 4000 kcal/week through exercise

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Lipid levels | Day 1 & 2 and Day 28 & 29 of each treatment phase
Postprandial glucose response | During week 1 and week 4 of each treatment phase
Fasting Insulin | Day 1 & 2 and Day 28 & 29 of each treatment phase
Insulin homeostasis modeling assessment | Day 1 & 2 and Day 28 & 29 of each treatment phase
Energy expenditure | During week 1 and week 4 of each treatment phase
body composition | Day 1 and Day 29 of each treatment phase
Antioxidant status | Day 1 & 2 and Day 28 & 29 of each treatment phase
Postprandial substrate utilization
Postprandial dietary fatty acid oxidation

CONTACTS AND LOCATIONS:
Overall Officials: Peter J.H. Jones, PhD, Principal Investigator — University of Manitoba - Richardson Centre for Functional Foods and Nutraceuticals
Locations (1):
- University of Manitoba - Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada